CLINICAL TRIAL: NCT02188069
Title: Canadian Spontaneous Coronary Artery Dissection (SCAD) Cohort Study
Brief Title: Canadian SCAD Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cardiology Research UBC (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jacqueline Saw, MD, Director of Research, Cardiology Research UBC
Other Study IDs: H14-00968
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Spontaneous Coronary Artery Dissection
Keywords: Non-atherosclerotic Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
SCAD (Spontaneous coronary artery dissection - tear in the arterial wall that is not related to trauma) is an under-diagnosed and poorly understood condition that mostly affects young women without common cardiovascular risk factors, and can result in heart attack and death. This observational study is designed to capture the disease's natural history and predisposing arteriopathies (medical conditions resulting in changes in the arteries), treatment strategies, long-term cardiovascular outcomes. It will also improve the diagnosis of SCAD on coronary angiography by participating clinicians, and provide guidance on investigating predisposing conditions.

DETAILED DESCRIPTION:
Background:

Spontaneous coronary artery dissection (SCAD) is an under-diagnosed and poorly understood condition that frequently affects young women without conventional cardiovascular (CV) risk factors, and can result in myocardial infarction (MI), cardiac arrest, and death. This condition has been inadequately researched, with no prospective studies evaluating management strategies, assessing the presence and impact of predisposing and precipitating causes, or assessing its effects on short- and long-term CV prognosis. Furthermore, many people presenting with MI due to SCAD have been mis-diagnosed due to the limitations of the current "gold-standard" diagnostic test (coronary angiography) for this condition, resulting in erroneous diagnoses such as atherosclerosis, microvascular dysfunction, Takotsubo cardiomyopathy, coronary artery spasm, or "normal" coronary arteries. As such, clinicians are uncertain about how to diagnose, investigate and manage patients with SCAD, and similarly, patients are uncertain about how this condition will affect their subsequent lifestyle and long-term cardiac prognosis. Therefore, we propose a large prospective multicenter Canadian SCAD cohort study to ascertain the natural history according to predisposing arteriopathies and treatment strategy on long-term CV outcomes. The design of this study will secondarily improve the diagnosis of SCAD on coronary angiography by participating clinicians, and provide guidance on investigating predisposing conditions.

Preliminary Data:

We have enrolled 170 NA-SCAD patients in our registry at Vancouver General Hospital. We discovered a very strong association between NA-SCAD and fibromuscular dysplasia (FMD), with ~80% of these NA-SCAD patients diagnosed with concomitant FMD. Of patients who underwent coronary angioplasty/stenting, successful and durable results occurred in only 33%. Of patients treated medically, those who had repeat coronary angiograms all showed angiographic healing.

Primary Objective:

1. To evaluate the overall natural history of NA-SCAD: (a) the overall in-hospital and long-term CV outcomes with NA-SCAD, (b) the prevalence and effects of predisposing arteriopathies on in-hospital and long-term CV outcomes, (c) the prevalence and impact of precipitating stressors on in-hospital and long-term CV events.

   Secondary Objectives:
2. To evaluate the in-hospital and long-term outcomes of conservative therapy and revascularization in patients with NA-SCAD.
3. To evaluate the presenting angiographic patterns of NA-SCAD.
4. To assess the incidence of spontaneous arterial healing with conservative medical therapy alone in NA-SCAD patients undergoing repeat angiography.

Hypotheses:

1. We hypothesize that NA-SCAD patients have a high risk of long-term recurrent CV events and FMD, as the most frequently observed predisposing condition confers lower subsequent risk compared to other arteriopathies, such as peripartum SCAD, with regards to CV outcomes. We hypothesize that precipitating stressors are common preceding the SCAD event in >50% of cases.
2. We hypothesize that NA-SCAD patients have a high risk of long-term CV events, and that patients who undergo revascularization have worse CV outcomes.
3. We hypothesize that the most common angiographic NA-SCAD pattern is diffuse stenosis.
4. We hypothesize that conservative medical therapy is associated with high rates of spontaneous healing.

Methodology:

Prospective Canadian observational cohort study enrolling 750 consecutive patients presenting with MI (NSTEMI or STEMI) due to NA-SCAD. Both women and men will be included. Rigorous coronary angiographic criteria with supplementary intracoronary imaging (reviewed by core laboratory) will be used for SCAD diagnosis. Detailed baseline demographics, targeted history for predisposing and precipitating factors, and screening laboratory tests will be performed. Patients will be prospectively followed for 3 years for CV events.

Significance:

This study will have significant impacts on the diagnosis, investigation, and management of NA-SCAD. Our diagnostic algorithm will help establish guidelines on SCAD diagnosis on coronary angiogram, which is currently elusive. Our rigorous clinical and laboratory screening will elucidate the prevalence of predisposing arteriopathies, which will help establish guidelines on investigation of SCAD patients. Knowledge of CV outcomes and natural history of NA-SCAD, especially stratified to predisposing arteriopathies, will establish prognosis, risk stratification, and management guidelines.

Knowledge Translation:

Our results will be disseminated to clinicians and patients through publications in scientific journals, physician scientific presentations, Healthy Heart Programs, patient educational sessions, educational website, and public media. Results from this study will help establish national and international guidelines on the diagnosis, investigation and management of NA-SCAD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted with troponin-positive ACS (NSTEMI or STEMI)
2. Documented NA-SCAD on coronary angiogram (including diagnosis with OCT or IVUS)

Exclusion Criteria:

1. Patients with troponin-negative ACS
2. Patients with typical atherosclerotic coronary artery disease in other coronary arterial segments with diameter stenosis ≥50%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective patients presenting with Spontaneous coronary artery dissection (SCAD)
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2014-06; Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Composite in-hospital outcome | During index admission
  Composite of all-cause mortality, stroke, reinfarction (31), cardiogenic shock (requiring medical or mechanical hemodynamic support), congestive heart failure, severe ventricular arrhythmia (requiring defibrillation or antiarrhythmic agents), repeat revascularization (or unplanned revascularization), and cardiac transplantation, collectively termed in-hospital major adverse events (MAE)
Composite follow-up outcome | 3 years post index event
  Composite of all-cause mortality, stroke, recurrent MI (including recurrent dissection), congestive heart failure and repeat revascularization, collectively termed major adverse cardiac events (MACE).

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Saw, MD, Principal Investigator — Vancouver General Hospital, University of British Columbia
Locations (20):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States
- Canada (19):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint Boniface General Hospital, Winnipeg, Manitoba
  - Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences General Site, Hamilton, Ontario
  - Saint Mary's, Kitchener, Ontario
  - London Health Sciences, London, Ontario
  - Southlake Regional Hospital, Newmarket, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Rough Valley Health System, Scarborough Village, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Health Centre (CUSM), Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - University of Montreal (CHUM), Montreal, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Saw J. Coronary angiogram classification of spontaneous coronary artery dissection. Catheter Cardiovasc Interv. 2014 Dec 1;84(7):1115-22. doi: 10.1002/ccd.25293. Epub 2013 Dec 4. PMID 24227590
- [Background] Saw J, Poulter R, Fung A, Wood D, Hamburger J, Buller CE. Spontaneous coronary artery dissection in patients with fibromuscular dysplasia: a case series. Circ Cardiovasc Interv. 2012 Feb 1;5(1):134-7. doi: 10.1161/CIRCINTERVENTIONS.111.966630. No abstract available. PMID 22338003
- [Background] Saw J, Ricci D, Starovoytov A, Fox R, Buller CE. Spontaneous coronary artery dissection: prevalence of predisposing conditions including fibromuscular dysplasia in a tertiary center cohort. JACC Cardiovasc Interv. 2013 Jan;6(1):44-52. doi: 10.1016/j.jcin.2012.08.017. Epub 2012 Dec 19. PMID 23266235
- [Background] Saw J, Aymong E, Mancini GB, Sedlak T, Starovoytov A, Ricci D. Nonatherosclerotic coronary artery disease in young women. Can J Cardiol. 2014 Jul;30(7):814-9. doi: 10.1016/j.cjca.2014.01.011. Epub 2014 Jan 23. PMID 24726091